CLINICAL TRIAL: NCT03842904
Title: A Randomised, Open Label 2-Way Cross-over Study to Compare the Effects of Inhaled Beclometasone/Formoterol/Glycopyrronium (TRIMBOW) pMDI to Beclometasone/Formoterol (FOSTAIR) pMDI on Hyperinflation and Expiratory Flow Limitation in Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study Comparing the Effects of Trimbow to Fostair in COPD
Acronym: TRIFLOW
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medicines Evaluation Unit Ltd (Industry)
Collaborators: Chiesi UK (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MEU 17/361; 2018-003113-17 (EudraCT Number)
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This is a phase IV, open-label, randomised, single centre, 2-way crossover study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trimbow pMDI (Experimental): Trimbow 87 micrograms/5 micrograms/9 micrograms pressurised inhalation solution.
  Interventions: Drug: Trimbow pMDI
- Fostair pMDI (Active Comparator): Fostair 100/6 micrograms per actuation pressurised inhalation solution.
  Interventions: Drug: Fostair pMDI

INTERVENTIONS:
Drug: Trimbow pMDI — Clinical Trial of an Investigational Medicinal Product (CTIMP)
  Arms: Trimbow pMDI
Drug: Fostair pMDI — Clinical Trial of an Investigational Medicinal Product (CTIMP)
  Arms: Fostair pMDI

SUMMARY:
A randomised, open label 2-way cross-over study to compare the effects of inhaled Beclometasone/Formoterol/Glycopyrronium (TRIMBOW) pMDI to Beclometasone/Formoterol (FOSTAIR) pMDI on hyperinflation and expiratory flow limitation in moderate to severe chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
This study will investigate the contributions of extra-fine glycopyrronium and formoterol (within triple therapy) to improvements in small airway function in COPD patients. This will be achieved by recruiting patients with hyperinflation, and measuring improvements in hyperinflation and expiratory flow limitation as measurements of small airway disease.

This study will help understand the mechanisms of action of the bronchodilators within BDP/FF/GB, and potentially encourage treatment of small airway disease in COPD with extra-fine bronchodilator treatments. This trial will be conducted in compliance with the Declaration of Helsinki (1964 and amendments) current Good Clinical Practices and all other applicable laws and regulations.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged 40 to 75 years with written informed consent obtained prior to any study-related procedure.
2. COPD diagnosis: Subjects with a diagnosis of moderate to severe COPD according to the GOLD 2018 COPD recommendations, with symptoms compatible with COPD for at least 1 year prior to screening.
3. Clinically stable COPD in the 6 weeks prior to screening and during the run-in period prior to randomisation.
4. Body mass index (BMI) in the range of 18.0 to 33.0 kg/m2 and with a minimum weight of 50 kg at screening.
5. Current smokers or ex-smokers with a smoking history of at least 10 pack years [pack-years = (number of cigarettes per day x number of years)/20].
6. A post-bronchodilator FEV1 ≥ 30 % and ≤ 70% of the predicted normal value and a post-bronchodilator FEV1/FVC ratio < 0.7 at screening.
7. Evidence of pre-bronchodilator hyperinflation (RV>120% predicted) at screening (V1) and baseline (V2).
8. Subject is willing and, in the opinion of the Investigator, able to change current COPD therapy as required by the protocol.
9. Subject is treated with double or triple therapy for at least 1 month prior to screening visit with either:

   1. Inhaled corticosteroids/long-acting β2-agonist, combination treatment (fixed and/or free)
   2. Inhaled corticosteroids and long-acting muscarinic antagonist
   3. inhaled corticosteroids/long-acting β2-agonist/long-acting muscarinic antagonist, combination treatment (fixed and/or free) In addition to the above subjects may be currently taking inhaled short acting β2-agonists and/or inhaled short acting anticholinergics.
10. A cooperative attitude and ability to be trained to correctly use the pMDI inhaler.
11. Compliance with inhaled Beclometasone run-in medication of between 80 to 120% at Visit 2 (baseline visit) and Visit 3 (Treatment Period 1, Day 1)

Exclusion Criteria:

1. Inability to comply with study procedures, required restrictions, study treatment intake or any other reason that the Investigator considers makes the patient unsuitable to participate.
2. COPD exacerbation requiring oral steroids and/or antibiotics, in the 8 weeks prior to screening or prior to randomisation.
3. Use of antibiotics for a respiratory tract infection in the 8 weeks prior to screening or prior to randomisation.
4. Inability to perform technically acceptable impulse oscillometry, whole body plethysmography or spirometry at screening, (V1) or baseline (V2).
5. Pregnant, lactating or breastfeeding women at screening, baseline or prior to randomisation. Positive urine pregnancy test at screening, baseline or prior to randomisation.
6. A history of one or more hospitalisations for COPD in the 12 months prior to screening or prior to randomisation.
7. Requires oxygen therapy, even on an occasional basis.
8. Known respiratory disorders other than COPD which may impact the efficacy or the safety of the study drug according to investigator's judgement. This can include but is not limited to known alpha-1 antitrypsin deficiency, active tuberculosis, lung cancer and bronchial carcinoma, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension and interstitial lung disease.
9. An abnormal and clinically significant 12-lead ECG which may impact the safety of the patient according to investigator's judgement.

   N.B: Subject whose electrocardiogram (ECG) (12 lead) shows QTcF>450 males or QTcF> 470 ms for females at screening are not eligible.
10. Medical diagnosis of narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that in the opinion of the investigator would prevent use of anticholinergic agents.
11. History of hypersensitivity to anticholinergics, β2-agonist, corticosteroids or any of the excipients contained in any of the formulations used in the trial which may raise contra-indications or impact the efficacy of the study drug according to the investigator's judgement.
12. Clinically significant laboratory abnormalities at screening indicating a significant or unstable concomitant disease which may impact the efficacy of the study drug or the safety of the patient, according to investigator's judgement.
13. Subjects with a history of chronic uncontrolled disease including, but not limited to, endocrine, active hyperthyroidism, neurological, hepatic, gastrointestinal, renal, haematological, urological, immunological, or ophthalmic diseases that the Investigator believes are clinically significant.
14. Uncontrolled cardiovascular disease: arrhythmias, angina, recent or suspected myocardial infarction, congestive heart failure, a history of unstable, or uncontrolled hypertension, or has been diagnosed with hypertension in the 3 months prior to screening or randomisation.
15. History of alcohol abuse and/or substance/drug abuse within 2 years prior to screening visit.
16. Has had major surgery, (requiring general anaesthesia) in the 8 weeks prior to screening or prior to randomisation, or has planned surgery through the end of the study.
17. Previous lung resection or lung reduction surgery.
18. Participation in another clinical trial and received investigational drug within 30 days (or 5 half-lives whichever is longer). N.B.: For biologic products with slow elimination a washout of at least 6 months needs to be met prior to screening visit.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Forced Expired Volume in 1 second (FEV1), L. | Pre-dose Day 1 and Day 5 (treatment period 1 & 2 - pre-dose, 30 minutes, 1, 2, 4, 6, 8, 10 and 12 hours post dose)
  To compare the effect of Trimbow and Fostair on FEV1 [(forced expiratory volume in 1 sec - changes from pre-dose day 1)].
Residual Volume (RV), L. | Pre-dose Day 1 and Day 5 (treatment period 1 & 2 - pre-dose, 1, 2, 4, 8 and 12 hours post dose)
  To compare the effect of Trimbow and Fostair on RV [(residual volume) - changes from pre-dose day 1)].

SECONDARY OUTCOMES:
Peripheral Respiratory Resistance (R5-R20), kPa/L/s. | Pre-dose Day 1 and Day 5 (treatment period 1 & 2 - pre-dose, 30 mins, 1, 2, 4, 6, 8, 10 & 12 hrs post dose)
  Impulse Oscillometry measurement
Expiratory Flow Limitation (Delta X5), kPa/L/s. | Pre-dose Day 1 and Day 5 (treatment period 1 & 2 - pre-dose, 30 mins, 1, 2, 4, 6, 8, 10 & 12 hrs post dose)
  Impulse Oscillometry measurement
Forced Vital Capacity (FVC), L | Baseline, Pre-dose Day 1 and Day 5 (treatment period 1 & 2 - pre-dose, 30 mins, 1, 2, 4, 6, 8, 10 & 12 hrs post dose)
  Spirometry measurement
Forced Expiratory Flow between 25-75% of FVC (FEF25-75%), L/s | Baseline, Pre-dose Day 1 and Day 5 (treatment period 1 & 2 - pre-dose, 30 mins, 1, 2, 4, 6, 8, 10 & 12 hrs post dose)
  Spirometry measurement
Resistance at 5Hz (R5), kPa/L/s | Baseline, Pre-dose Day 1 and Day 5 (treatment period 1 & 2 - pre-dose, 30 mins, 1, 2, 4, 6, 8, 10 & 12 hrs post dose)
  Impulse Oscillometry measurement
Reactance at 5Hz (X5), kPa/L/s | Baseline, Pre-dose Day 1 and Day 5 (treatment period 1 & 2 - pre-dose, 30 mins, 1, 2, 4, 6, 8, 10 & 12 hrs post dose)
  Impulse Oscillometry measurement
Resonance Frequency (Fres), Hz | Baseline, Pre-dose Day 1 and Day 5 (treatment period 1 & 2 - pre-dose, 30 mins, 1, 2, 4, 6, 8, 10 & 12 hrs post dose)
  Impulse Oscillometry measurement
Reactance Area (AX), kPa/L | Baseline, Pre-dose Day 1 and Day 5 (treatment period 1 & 2 - pre-dose, 30 mins, 1, 2, 4, 6, 8, 10 & 12 hrs post dose)
  Impulse Oscillometry measurement
Total Lung Capacity (TLC), L | Baseline, Pre-dose Day 1 and Day 5 (treatment period 1 & 2 - pre-dose, 1, 2, 4, 8 & 12 hrs post dose)
  Plethysmography measurement
Functional Residual Capacity (FRC), L | Baseline, Pre-dose Day 1 and Day 5 (treatment period 1 & 2 - pre-dose, 1, 2, 4, 8 & 12 hrs post dose)
  Plethysmography measurement
Inspiratory Capacity (IC), L | Baseline, Pre-dose Day 1 and Day 5 (treatment period 1 & 2 - pre-dose, 1, 2, 4, 8 & 12 hrs post dose)
  Plethysmography measurement
Specific Airway Conductance (SGaw), L/s/kPa/L | Baseline, Pre-dose Day 1 and Day 5 (treatment period 1 & 2 - pre-dose, 1, 2, 4, 8 & 12 hrs post dose)
  Plethysmography measurement
Airway Resistance (Raw), kPa/L/s | Baseline, Pre-dose Day 1 and Day 5 (treatment period 1 & 2 - pre-dose, 1, 2, 4, 8 & 12 hrs post dose)
  Plethysmography measurement
Forced Expired Volume in 1 second (FEV1), L. | Baseline and Day 5 (treatment period 1 & 2 - pre-dose, 30 mins, 1, 2, 4, 6, 8, 10 & 12 hrs post dose)
  Spirometry measurement
Residual Volume (RV), L. | Baseline and Day 5 (treatment period 1 & 2 - pre-dose, 1, 2, 4, 8 & 12 hrs post dose)
  Plethysmography measurement

OTHER OUTCOMES:
Frequency of AEs reported | From consent through study completion (study duration is approx. 5-10 weeks)
  To assess the safety and tolerability of the study treatment, as frequency of AEs reported.

CONTACTS AND LOCATIONS:
Overall Officials: David Rogers, Study Director — Medicines Evaluation Unit Ltd
Locations (1):
- The Medicines Evaluation Unit (MEU), Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dean J, Panainte C, Khan N, Singh D. The TRIFLOW study: a randomised, cross-over study evaluating the effects of extrafine beclometasone/formoterol/glycopyrronium on gas trapping in COPD. Respir Res. 2020 Dec 9;21(1):323. doi: 10.1186/s12931-020-01589-5. PMID 33298062
- See also: Research facility website — http://www.meu.org.uk/